CLINICAL TRIAL: NCT01391286
Title: A Multicenter, Double-masked, Randomized, Parallel-group Study Assessing the Safety and Efficacy of Once-daily Application of Bimatoprost Solution 0.03% Compared to Vehicle to Treat Chemotherapy-induced Hypotrichosis of the Eyelashes in Japanese Subjects
Brief Title: Safety and Efficacy Study of Bimatoprost in Japanese Patients With Chemotherapy-Induced Eyelash Hypotrichosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 192024-067
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Results first posted 2013-07-09 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-04

CONDITIONS: Eyelash Hypotrichosis
MeSH Terms: interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bimatoprost solution 0.03% (Experimental): One drop of bimatoprost solution 0.03% applied along each upper eyelid margin once daily in the evening for 4 months.
  Interventions: Drug: bimatoprost solution 0.03%
- bimatoprost vehicle solution (Placebo Comparator): One drop of bimatoprost vehicle solution applied along each upper eyelid margin once daily in the evening for 4 months.
  Interventions: Drug: bimatoprost vehicle solution

INTERVENTIONS:
Drug: bimatoprost solution 0.03% — One drop of bimatoprost solution 0.03% applied along each upper eyelid margin once daily in the evening for 4 months.
  Other Names: LATISSE®
  Arms: bimatoprost solution 0.03%
Drug: bimatoprost vehicle solution — One drop of bimatoprost vehicle solution applied along each upper eyelid margin once daily in the evening for 4 months.
  Arms: bimatoprost vehicle solution

SUMMARY:
This study will evaluate the safety and efficacy of bimatoprost solution 0.03% compared with vehicle in Japanese adults with hypotrichosis of the eyelashes following chemotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have inadequate eyelashes due to chemotherapy treatment
* Treated for solid tumors such as breast or colorectal cancer in early stages where the cancer has not spread outside the primary organ (eg, stage 1, 2 or 3a for breast cancer)
* Have completed chemotherapy treatment for at least 4 weeks but not more than 24 weeks and all side effects related to chemotherapy are recovered, improved or maintained, with the exception of hair loss

Exclusion Criteria:

* Any disease/infection/abnormality of the eye or area around the eye
* Any ocular surgery within 3 months or anticipated need for ocular surgery during the study
* Any permanent eyeliner or implants of any kind or anticipated use of false eyelashes
* Any semi-permanent eyelash tint, dye, curl or eyelash extension application within 3 months
* Use of any over-the-counter eyelash growth product within 6 months or any use of prescription eyelash growth products
* Use of treatments which may affect hair growth (eg, minoxidil) within 6 months except for prior chemotherapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2012-05-25 (Actual); Study Completion 2012-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Chiba, Japan

REFERENCES:
- [Background] Harii K, Arase S, Tsuboi R, Weng E, Daniels S, VanDenburgh A. Bimatoprost for eyelash growth in Japanese subjects: two multicenter controlled studies. Aesthetic Plast Surg. 2014 Apr;38(2):451-60. doi: 10.1007/s00266-014-0293-7. Epub 2014 Mar 19. PMID 24643895

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost Solution 0.03% | Bimatoprost Vehicle Solution
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost Solution 0.03% | Bimatoprost Vehicle Solution | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Customized [Number; unit: Participants]
  < 45 Years | 8 | 3 | 11
  45 to 65 Years | 10 | 12 | 22
  > 65 Years | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least a 1-Grade Increase in Overall Eyelash Prominence Using the Global Eyelash Assessment Scale (GEA)
Description: The investigator evaluated the patient's eyelash prominence using the GEA 4-point scale: 1= minimal, 2= moderate, 3= marked and 4= very marked at Baseline and Month 4. At least a 1-grade increase in the GEA score from Baseline indicated improvement.
Time Frame: Baseline, Month 4
Population: Intent to treat population included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Bimatoprost Solution 0.03% | Bimatoprost Vehicle Solution
Number analyzed (Participants) | 18 | 18
Percentage of participants | 88.9 | 27.8

2. Secondary Outcome: Change From Baseline in Eyelash Length as Measured by Digital Image Analysis (DIA)
Description: Photographs were taken of the eyelashes and assessed using DIA. Length was measured in millimeters (mm). Data from both eyes were averaged for each participant for analysis. A positive change from Baseline indicated longer length (improvement).
Time Frame: Baseline, Month 4
Population: Participants from the Intent to treat population with data available for analysis.
Measure: Median (Full Range); unit: mm
Arm/Group | Bimatoprost Solution 0.03% | Bimatoprost Vehicle Solution
Number analyzed (Participants) | 17 | 17
mm
  Baseline | 5.70 (1.397) [2.5 to 7.3] | 5.00 (1.543) [1.4 to 7.2]
  Change from Baseline at Month 4 | 2.70 (1.574) [0.6 to 6.3] | 0.6 (1.317) [-0.6 to 3.3]

3. Secondary Outcome: Change From Baseline in Eyelash Thickness as Measured by DIA
Description: Photographs were taken of the eyelashes and assessed using DIA. Eyelash thickness (fullness) was assessed across both eyes as an average and is measured in millimeters squared (mm^2). A positive change from Baseline indicated fuller eyelashes (improvement).
Time Frame: Baseline, Month 4
Population: Participants from the Intent to treat population with data available for analysis.
Measure: Median (Full Range); unit: mm^2
Arm/Group | Bimatoprost Solution 0.03% | Bimatoprost Vehicle Solution
Number analyzed (Participants) | 15 | 14
mm^2
  Baseline | 0.60 (0.456) [0.1 to 1.5] | 0.45 (0.294) [0.1 to 1.1]
  Change from Baseline at Month 4 | 0.80 (0.460) [0.1 to 2.0] | 0.25 (0.393) [-0.2 to 0.9]

4. Secondary Outcome: Change From Baseline in Eyelash Darkness as Measured by DIA
Description: Photographs were taken of the eyelashes and assessed using DIA. Eyelash darkness was measured in both eyes and averaged for analysis using a scale where 0=black and 255=white. A negative change from Baseline indicated darker eyelashes (improvement).
Time Frame: Baseline, Month 4
Population: Participants from the Intent to treat population with data available for analysis.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Bimatoprost Solution 0.03% | Bimatoprost Vehicle Solution
Number analyzed (Participants) | 15 | 14
Units on a scale
  Baseline | 140.15 (21.855) [98.7 to 173.7] | 144.98 (18.561) [123.8 to 181.4]
  Change from Baseline at Month 4 | -19.40 (12.666) [-53.4 to 3.0] | -10.03 (18.248) [-23.5 to 33.6]

ADVERSE EVENTS:
Arm/Group | Bimatoprost Solution 0.03% | Bimatoprost Vehicle Solution
Serious Adverse Events (participants affected / at risk) | 0/18 | 2/18
Other Adverse Events (participants affected / at risk) | 12/18 | 13/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost Solution 0.03% (N=18) | Bimatoprost Vehicle Solution (N=18)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost Solution 0.03% (N=18) | Bimatoprost Vehicle Solution (N=18)
Hypothyroidism (Endocrine disorders) | 0 | 1
Eye pruritus (Eye disorders) | 1 | 1
Erythema of eyelid (Eye disorders) | 1 | 0
Blepharitis (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Periodontitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Sensation of pressure (General disorders) | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 4
Cellulitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 4 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Affective disorder (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Pruritus genital (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Milia (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 0
Blood pressure fluctuation (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.